CLINICAL TRIAL: NCT02469077
Title: Reduced Opioid Analgesic Requirements Via Improved Endogenous Opioid Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Stephen Bruehl, PhD, Professor of Anesthesiology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 141862; R01DA037891 (NIH)
Record Dates: First submitted 2015-05-07; First posted 2015-06-11 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Chronic Pain
Keywords: Chronic Low Back Pain
MeSH Terms: conditions — Chronic Pain | interventions — Morphine; Naloxone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 6 week aerobic exercise intervention (Experimental): Participants randomly assigned to the exercise condition will complete an 18 session aerobic exercise manipulation supervised by an American College of Sports Medicine-certified personal trainer (3 exercise sessions per week for 6 weeks). Immediately before and after participating in this intervention arm, participants will undergo laboratory evoked thermal pain response testing with placebo-controlled morphine and naloxone administration to assess mechanisms of exercise-related changes.
  Interventions: Behavioral: 6 week aerobic exercise intervention; Drug: Placebo; Drug: Morphine; Drug: naloxone
- Normal exercise (control) (Active Comparator): Participants assigned to the control condition will not undergo any exercise manipulation during this 6 week period, and will be asked to continue their current activity levels and not engage in any additional exercise activity during the study period. Immediately before and after participating in this intervention arm, participants will undergo laboratory evoked thermal pain response testing with placebo-controlled morphine and naloxone administration to assess mechanisms of exercise-related changes.
  Interventions: Drug: Placebo; Drug: Morphine; Drug: naloxone

INTERVENTIONS:
Behavioral: 6 week aerobic exercise intervention — Participants randomly assigned to the 6 week aerobic exercise intervention will complete an 18 session aerobic exercise manipulation supervised by an American College of Sports Medicine-certified personal trainer (3 exercise sessions per week for 6 weeks).
  Each exercise session will consist of a 5 minute warm-up, 30 minutes of aerobic exercise, followed by a 5 minute cool-down period. Aerobic exercise will consist of treadmill walking/running, stepping, elliptical, or cycling exercise as preferred by the participant. Duration of exercise will be standardized at 30 minutes with a target exercise intensity between 70-85% Heart Rate Reserve (RPE = 15, hard). Because of the focus on de-conditioned individuals with Chronic Low Back Pain, the duration and intensity of exercise will be progressively increased up to target during the first two weeks to avoid symptom exacerbation and minimize study drop-out.
  Arms: 6 week aerobic exercise intervention
Drug: Placebo — In randomized order (crossover) across 3 laboratory sessions each approximately 5 days apart, participants will undergo laboratory evoked thermal pain response testing with: 1) 4 doses of saline placebo (20ml each), 2) an 8mg dose of naloxone (in 20ml saline vehicle), followed by saline, 4mg naloxone, and saline, or 3) morphine sulfate (0.03 mg/kg in 20ml saline vehicle initially, followed by 3 incremental doses of 0.02mg/kg each).
  Other Names: normal saline placebo
Drug: Morphine — In randomized order (crossover) across 3 laboratory sessions each approximately 5 days apart, participants will undergo laboratory evoked thermal pain response testing with: 1) 4 doses of saline placebo (20ml each), 2) an 8mg dose of naloxone (in 20ml saline vehicle), followed by saline, 4mg naloxone, and saline, or 3) morphine sulfate (0.03 mg/kg in 20ml saline vehicle initially, followed by 3 incremental doses of 0.02mg/kg each).
  Other Names: Astramorph
Drug: naloxone — In randomized order (crossover) across 3 laboratory sessions each approximately 5 days apart, participants will undergo laboratory evoked thermal pain response testing with: 1) 4 doses of saline placebo (20ml each), 2) an 8mg dose of naloxone (in 20ml saline vehicle), followed by saline, 4mg naloxone, and saline, or 3) morphine sulfate (0.03 mg/kg in 20ml saline vehicle initially, followed by 3 incremental doses of 0.02mg/kg each).
  Other Names: narcan

SUMMARY:
Chronic Pain (CP) management has increasingly utilized long-term opioid analgesic therapy, a change associated with increased opioid abuse (via greater exposure in vulnerable individuals), non-pain health consequences (hormone changes, falls), and a dramatic rise in opioid-related overdoses and deaths. Treatment strategies that minimize the need for chronic high-dose opioids are sorely needed. This project will test the novel hypothesis that effective pain relief can be achieved at lower opioid analgesic doses by increasing levels of endogenous opioids (EOs).

DETAILED DESCRIPTION:
There are three separate goals of the study: 1) test the effects of the intervention (versus control) on clinical outcomes, 2) test for endogenous opioid mechanisms of the intervention (indexed by the difference in laboratory evoked pain response between placebo and naloxone drug conditions), and 3) test the effects of the intervention on morphine responses (indexed by the difference in evoked pain response between placebo and morphine laboratory drug conditions).

This project will determine whether enhancing endogenous opioids (via aerobic exercise training) permits achieving desired levels of analgesia with lower dosages of opioid analgesics, and fewer side effects and abuse-relevant drug effects. This 4 year project will test study hypotheses in a sample of 116 chronic low back pain patients. The study will have two key elements: 1) a randomized, controlled aerobic exercise manipulation in CP patients completing daily electronic pain diaries and 2) laboratory evoked thermal pain protocols pre- and post-exercise permitting direct examination of changes in both opioid analgesic effects (in response to a series of incremental morphine doses) and EO activity (indexed by comparing pain responses after placebo vs. opioid blockade).

The study will use a 6 week supervised aerobic exercise manipulation, with subjects randomly assigned to the exercise protocol or a no exercise control condition.

The study will employ a mixed between/within-subjects design using double-blind, counterbalanced, placebo-controlled administration of both an opioid antagonist (naloxone) and an opioid agonist (morphine). All participants will undergo three identical laboratory pain-induction sessions (each ≈5 days apart) prior to randomization to experimental condition, and again at the end of the 6 week exercise manipulation period (regardless of exercise group assignment) during which they will receive the 3 study drugs and participate in controlled laboratory evaluation of evoked thermal pain responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Intact cognitive status and ability to provide informed consent
* Ability to read and write in English sufficiently to understand and complete study questionnaires
* Age 18-55 inclusive
* Presence of persistent daily low back pain of at least three months duration and of at least a 3/10 in average intensity

Exclusion Criteria:

* Engagement in > 2 days/wk and > 60 min/wk of moderate or vigorous intensity activity based on responses to 6 validated survey questions at screening (CDC BRFSS)
* History of renal or hepatic dysfunction
* Current or past alcohol or substance dependence
* A history of PTSD, psychotic, or bipolar disorders
* Chronic pain due to malignancy (e.g., cancer), autoimmune disorders (e.g., rheumatoid arthritis, lupus), or fibromyalgia
* Recent daily opiate use
* Use of any opioid analgesic medications within 72 hours of study participation (confirmed through rapid urine screening conducted prior to study participation)
* Females who are pregnant
* History of cardiovascular disease (including myocardial infarction)
* History of seizure disorder
* Prior allergic reaction/intolerance to morphine or its analogs
* Presence of cardiac disease or any other medical condition that would make engaging in the aerobic exercise manipulation unsafe

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2015-08; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bruehl, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Rush University, Chicago, Illinois
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bement MK, Sluka KA. Low-intensity exercise reverses chronic muscle pain in the rat in a naloxone-dependent manner. Arch Phys Med Rehabil. 2005 Sep;86(9):1736-40. doi: 10.1016/j.apmr.2005.03.029. PMID 16181935
- [Background] Bruehl S, Burns JW, Gupta R, Buvanendran A, Chont M, Kinner E, Schuster E, Passik S, France CR. Endogenous opioid function mediates the association between laboratory-evoked pain sensitivity and morphine analgesic responses. Pain. 2013 Sep;154(9):1856-1864. doi: 10.1016/j.pain.2013.06.002. Epub 2013 Jun 6. PMID 23748117
- [Background] Bruehl S, Burns JW, Gupta R, Buvanendran A, Chont M, Schuster E, France CR. Endogenous opioid inhibition of chronic low-back pain influences degree of back pain relief after morphine administration. Reg Anesth Pain Med. 2014 Mar-Apr;39(2):120-5. doi: 10.1097/AAP.0000000000000058. PMID 24553304
- [Background] Bruehl S, Chung OY, Burns JW, Biridepalli S. The association between anger expression and chronic pain intensity: evidence for partial mediation by endogenous opioid dysfunction. Pain. 2003 Dec;106(3):317-324. doi: 10.1016/S0304-3959(03)00319-1. PMID 14659514
- [Background] Chatzitheodorou D, Kabitsis C, Malliou P, Mougios V. A pilot study of the effects of high-intensity aerobic exercise versus passive interventions on pain, disability, psychological strain, and serum cortisol concentrations in people with chronic low back pain. Phys Ther. 2007 Mar;87(3):304-12. doi: 10.2522/ptj.20060080. Epub 2007 Feb 6. PMID 17284546
- [Background] Droste C, Meyer-Blankenburg H, Greenlee MW, Roskamm H. Effect of physical exercise on pain thresholds and plasma beta-endorphins in patients with silent and symptomatic myocardial ischaemia. Eur Heart J. 1988 Dec;9 Suppl N:25-33. doi: 10.1093/eurheartj/9.suppl_n.25. PMID 3246253
- [Background] Eriksson SV, Lundeberg T, Lundeberg S. Interaction of diazepam and naloxone on acupuncture induced pain relief. Am J Chin Med. 1991;19(1):1-7. doi: 10.1142/S0192415X91000028. PMID 1654741
- [Background] Ernst M, Lee MH. Influence of naloxone on electro-acupuncture analgesia using an experimental dental pain test. Review of possible mechanisms of action. Acupunct Electrother Res. 1987;12(1):5-22. doi: 10.3727/036012987816358940. PMID 2883837
- [Background] Fritz MS, Mackinnon DP. Required sample size to detect the mediated effect. Psychol Sci. 2007 Mar;18(3):233-9. doi: 10.1111/j.1467-9280.2007.01882.x. PMID 17444920
- [Background] Haier RJ, Quaid K, Mills JC. Naloxone alters pain perception after jogging. Psychiatry Res. 1981 Oct;5(2):231-2. doi: 10.1016/0165-1781(81)90052-4. No abstract available. PMID 6945616
- [Background] Hoffman MD, Shepanski MA, Mackenzie SP, Clifford PS. Experimentally induced pain perception is acutely reduced by aerobic exercise in people with chronic low back pain. J Rehabil Res Dev. 2005 Mar-Apr;42(2):183-90. doi: 10.1682/jrrd.2004.06.0065. PMID 15944883
- [Background] Hutchinson MR, Zhang Y, Shridhar M, Evans JH, Buchanan MM, Zhao TX, Slivka PF, Coats BD, Rezvani N, Wieseler J, Hughes TS, Landgraf KE, Chan S, Fong S, Phipps S, Falke JJ, Leinwand LA, Maier SF, Yin H, Rice KC, Watkins LR. Evidence that opioids may have toll-like receptor 4 and MD-2 effects. Brain Behav Immun. 2010 Jan;24(1):83-95. doi: 10.1016/j.bbi.2009.08.004. Epub 2009 Aug 11. PMID 19679181
- [Background] Janal MN, Colt EWD, Clark CW, Glusman M. Pain sensitivity, mood and plasma endocrine levels in man following long-distance running: effects of naloxone. Pain. 1984 May;19(1):13-25. doi: 10.1016/0304-3959(84)90061-7. PMID 6330643
- [Background] King CD, Goodin B, Kindler LL, Caudle RM, Edwards RR, Gravenstein N, Riley JL 3rd, Fillingim RB. Reduction of conditioned pain modulation in humans by naltrexone: an exploratory study of the effects of pain catastrophizing. J Behav Med. 2013 Jun;36(3):315-27. doi: 10.1007/s10865-012-9424-2. Epub 2012 Apr 26. PMID 22534819
- [Background] Koltyn KF. Analgesia following exercise: a review. Sports Med. 2000 Feb;29(2):85-98. doi: 10.2165/00007256-200029020-00002. PMID 10701712
- [Background] Meeus M, Roussel NA, Truijen S, Nijs J. Reduced pressure pain thresholds in response to exercise in chronic fatigue syndrome but not in chronic low back pain: an experimental study. J Rehabil Med. 2010 Oct;42(9):884-90. doi: 10.2340/16501977-0595. PMID 20878051
- [Background] Olausson B, Eriksson E, Ellmarker L, Rydenhag B, Shyu BC, Andersson SA. Effects of naloxone on dental pain threshold following muscle exercise and low frequency transcutaneous nerve stimulation: a comparative study in man. Acta Physiol Scand. 1986 Feb;126(2):299-305. doi: 10.1111/j.1748-1716.1986.tb07818.x. PMID 3486546
- [Background] Paulev PE, Thorboll JE, Nielsen U, Kruse P, Jordal R, Bach FW, Fenger M, Pokorski M. Opioid involvement in the perception of pain due to endurance exercise in trained man. Jpn J Physiol. 1989;39(1):67-74. doi: 10.2170/jjphysiol.39.67. PMID 2542682
- [Background] Preacher KJ, Hayes AF. SPSS and SAS procedures for estimating indirect effects in simple mediation models. Behav Res Methods Instrum Comput. 2004 Nov;36(4):717-31. doi: 10.3758/bf03206553. PMID 15641418
- [Background] Preacher KJ, Hayes AF. Asymptotic and resampling strategies for assessing and comparing indirect effects in multiple mediator models. Behav Res Methods. 2008 Aug;40(3):879-91. doi: 10.3758/brm.40.3.879. PMID 18697684
- [Background] Prentice RL. A generalization of the probit and logit methods for dose response curves. Biometrics. 1976 Dec;32(4):761-8. PMID 1009225
- [Background] Rainville J, Hartigan C, Jouve C, Martinez E. The influence of intense exercise-based physical therapy program on back pain anticipated before and induced by physical activities. Spine J. 2004 Mar-Apr;4(2):176-83. doi: 10.1016/j.spinee.2003.08.031. PMID 15016395
- [Background] Scheef L, Jankowski J, Daamen M, Weyer G, Klingenberg M, Renner J, Mueckter S, Schurmann B, Musshoff F, Wagner M, Schild HH, Zimmer A, Boecker H. An fMRI study on the acute effects of exercise on pain processing in trained athletes. Pain. 2012 Aug;153(8):1702-1714. doi: 10.1016/j.pain.2012.05.008. Epub 2012 Jun 16. PMID 22704853
- [Background] Shnayderman I, Katz-Leurer M. An aerobic walking programme versus muscle strengthening programme for chronic low back pain: a randomized controlled trial. Clin Rehabil. 2013 Mar;27(3):207-14. doi: 10.1177/0269215512453353. Epub 2012 Jul 31. PMID 22850802
- [Background] Stagg NJ, Mata HP, Ibrahim MM, Henriksen EJ, Porreca F, Vanderah TW, Philip Malan T Jr. Regular exercise reverses sensory hypersensitivity in a rat neuropathic pain model: role of endogenous opioids. Anesthesiology. 2011 Apr;114(4):940-8. doi: 10.1097/ALN.0b013e318210f880. PMID 21386701
- [Background] Sun Y, Gan TJ, Dubose JW, Habib AS. Acupuncture and related techniques for postoperative pain: a systematic review of randomized controlled trials. Br J Anaesth. 2008 Aug;101(2):151-60. doi: 10.1093/bja/aen146. Epub 2008 Jun 2. PMID 18522936
- [Background] Ulett GA, Han S, Han JS. Electroacupuncture: mechanisms and clinical application. Biol Psychiatry. 1998 Jul 15;44(2):129-38. doi: 10.1016/s0006-3223(97)00394-6. PMID 9646895
- [Background] Willer JC, Le Bars D, De Broucker T. Diffuse noxious inhibitory controls in man: involvement of an opioidergic link. Eur J Pharmacol. 1990 Jul 3;182(2):347-55. doi: 10.1016/0014-2999(90)90293-f. PMID 2168836
- [Derived] Bruehl S, Stone AL, Palmer C, Edwards DA, Buvanendran A, Gupta R, Chont M, Kennedy M, Burns JW. Self-reported cumulative medical opioid exposure and subjective responses on first use of opioids predict analgesic and subjective responses to placebo-controlled opioid administration. Reg Anesth Pain Med. 2019 Jan;44(1):92-99. doi: 10.1136/rapm-2018-000008. PMID 30640659

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 117 subjects consented and participated in Visit 1 to evaluate the nature of chronic back pain and confirm eligibility to engage in exercise manipulation. 15 subjects were discontinued from participation following this assessment. 9 additional subjects discontinued during preintervention lab session period.
Period: Pre Randomization - Pre Intervention
Arm/Group | 6 Week Aerobic Exercise Intervention | Normal Exercise (Control)
Started (Order of preexercise intervention placebo/morphine/naloxone randomizedeach subject) | 44 | 49
Pre Intervention Placebo | 44 | 49
Pre Intervention Morpine | 44 | 49
Pre Intervention Naloxone | 44 | 49
Completed | 44 | 49
Not Completed | 0 | 0
Period: Post Randomization/Intervention Period
Arm/Group | 6 Week Aerobic Exercise Intervention | Normal Exercise (Control)
Started | 44 | 49
Completed | 40 | 45
Not Completed | 4 | 4
Not completed — Scheduling issues | 3 | 2
Not completed — Relocated | 1 | 1
Not completed — Conflicting health issues | 0 | 1
Period: Post Intervention /Followup
Arm/Group | 6 Week Aerobic Exercise Intervention | Normal Exercise (Control)
Started (Order ofpostexercise intervention assessmentwith placebo/morphine/naloxone randomized foreachsubject) | 40 | 45
Post Intervention Placebo | 39 | 45
Post Intervention Morphine | 40 | 45
Post Intervention Naloxone | 39 | 44
Completed | 38 | 44
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Exercise Plus Placebo/Morphine/Naloxone: Participants randomly assigned to the exercise condition will complete an 18 session aerobic exercise manipulation supervised by an American College of Sports Medicine certified personal trainer (3 exercise sessions per week for 6 weeks). Immediately before and after participating in this intervention arm, participants will undergo the placebo-controlled morphine and naloxone administration intervention to assess mechanisms of exercise-related changes.
  exercise: Each exercise session will consist of a 5 minute warm-up, 30 minutes of aerobic exercise, followed by a 5 minute cool-down period. Aerobic exercise will consist of treadmill walking/running, stepping, elliptical, or cycling exercise as preferred by the participant. Duration of exercise will be standardized at 30 minutes with a target exercise intensity between 70-85% Heart Rate Reserve (RPE = 15, hard). Because of the focus on de-conditioned individuals with Chronic Low Back Pain, the duration and intensity of exercise wil
- Placebo/Morphine/Naloxone: Participants assigned to the control condition will not undergo any manipulation during this 6 week period, and will be asked to continue their current activity levels and not engage in any additional exercise activity during the study period. Immediately before and after participating in this intervention arm, participants will undergo the placebo-controlled morphine and naloxone administration intervention to assess mechanisms of exercise-related changes.
  Placebo: In randomized order (crossover) across 3 laboratory sessions each approximately 5 days apart, participants will receive: 1) 4 doses of saline placebo (20ml each), 2) an 8mg dose of naloxone (in 20ml saline vehicle), followed by saline, 4mg naloxone, and saline, or 3) morphine sulfate (0.03 mg/kg in 20ml saline vehicle initially, followed by 3 incremental doses of 0.02mg/kg each)
  Morphine: In randomized order (crossover) across 3 laboratory sessions each approximately 5 days apart, participants will receive: 1) 4 dose
- Total: Total of all reporting groups
Arm/Group | Exercise Plus Placebo/Morphine/Naloxone | Placebo/Morphine/Naloxone | Total
Number analyzed (Participants) | 38 | 44 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 44 | 82
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 28 | 48
  Male | 18 | 16 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 36 | 39 | 75
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 15 | 25
  White | 23 | 25 | 48
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 44 | 82

OUTCOME MEASURES:

1. Primary Outcome: Mean of the Change in Morphine Dosage (in mg) Required to Achieve 25% Reduction in Thermal Evoked Pain Responses Relative to Baseline (Pre-intervention) Placebo Condition Responses
Description: At a laboratory testing day pre and post intervention each participant received morphine sulphate (0.3mg/kg in 20ml saline vehicle initially, followed by 3 incremental doses of 0.02 mg/kg each with testing for thermal evoked pain response. Weight adjusted dosing was used by multiplying the weight of each patient in kg by 0.3mg (dose 1 only) or by .02mg (doses 2-4), with all doses infused in 20mL saline vehicle.
  Mean of the change in morphine dosage required to achieve 25 % reduction in thermal evoked pain responses on testing day at baseline (pre-intervention) and post intervention. Positive values for the change in the mean between pre and post intervention indicated decreased morphine requirements post intervention.
Time Frame: At pre-intervention baseline laboratory assessment and again post-intervention (an expected average of 6 weeks later)
Population: Data was not available for analysis of 2 participants in the exercise arm and 1 participant in the control arm
Measure: Mean (Standard Deviation); unit: mg
Groups:
- 6 Week Aerobic Exercise Intervention: Participants randomly assigned to the exercise condition will complete an 18 session aerobic exercise manipulation supervised by an American College of Sports Medicine-certified personal trainer (3 exercise sessions per week for 6 weeks). Immediately before and after participating in this intervention arm, participants will undergo the placebo-controlled morphine and naloxone administration intervention to assess mechanisms of exercise-related changes.
  exercise: Each exercise session will consist of a 5 minute warm-up, 30 minutes of aerobic exercise, followed by a 5 minute cool-down period. Aerobic exercise will consist of treadmill walking/running, stepping, elliptical, or cycling exercise as preferred by the participant. Duration of exercise will be standardized at 30 minutes with a target exercise intensity between 70-85% Heart Rate Reserve (RPE = 15, hard). Because of the focus on de-conditioned individuals with Chronic Low Back Pain, the duration and intensity of exercise wil
- Normal Exercise (Control): Participants assigned to the control condition will not undergo any manipulation during this 6 week period, and will be asked to continue their current activity levels and not engage in any additional exercise activity during the study period. Immediately before and after participating in this intervention arm, participants will undergo the placebo-controlled morphine and naloxone administration intervention to assess mechanisms of exercise-related changes.
  Placebo: In randomized order (crossover) across 3 laboratory sessions each approximately 5 days apart, participants will receive: 1) 4 doses of saline placebo (20ml each), 2) an 8mg dose of naloxone (in 20ml saline vehicle), followed by saline, 4mg naloxone, and saline, or 3) morphine sulfate (0.03 mg/kg in 20ml saline vehicle initially, followed by 3 incremental doses of 0.02mg/kg each)
  Morphine: In randomized order (crossover) across 3 laboratory sessions each approximately 5 days apart, participants will receive: 1) 4 dose
Arm/Group | 6 Week Aerobic Exercise Intervention | Normal Exercise (Control)
Number analyzed (Participants) | 36 | 43
mg
  Baseline (pre intervention) | 4.17 (1.82) | 6.34 (5.63)
  Change after 6 week intervention period | -1.62 (4.46) | 0.92 (5.16)
Statistical Analysis 1: Comparison: 6 Week Aerobic Exercise Intervention vs Normal Exercise (Control); Statistical analysis applies to change after 6 week intervention period; Test type: Superiority; p = 0.12, ANCOVA

2. Primary Outcome: Mean Change in 5-day Electronic Diary Ratings of Low Back Pain Intensity
Description: Mean change in 5-day electronic diary ratings of low back pain intensity from pre intervention baseline to post intervention. 9 point pain scale assessing pain intensity with 0 represents no pain and 8 represents worst possible pain. Positive values indicate reduced pain post intervention.
Time Frame: At pre-intervention baseline and again post-intervention (an expected average of 6 weeks later)
Population: Data was not available for analysis of 4 participants in the exercise arm and 11 participants in the control arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 6 Week Aerobic Exercise Intervention | Normal Exercise (Control)
Number analyzed (Participants) | 34 | 33
units on a scale
  Baseline (pre intervention) | 2.75 (1.20) | 2.82 (1.38)
  Change after 6 week intervention period | 0.72 (1.18) | 0.18 (0.91)
Statistical Analysis 1: Comparison: 6 Week Aerobic Exercise Intervention vs Normal Exercise (Control); Statistical analysis applies to change after 6 week intervention period; Test type: Superiority; p = .04, ANCOVA

3. Secondary Outcome: Mean Change in Placebo Condition Ratings of Acute Thermal Pain Intensity on the McGill Pain Questionnaire-Short Form
Description: Mean change in placebo condition ratings of acute thermal pain intensity using the McGill Pain Questionnaire-Short Form on 3 testing days at baseline (per intervention) and post intervention. The score ranges from 0-33 where 0 represents no pain and 33 represents most intense pain. Positive change values indicate decreased pain responsiveness post intervention.
Time Frame: At pre-intervention baseline laboratory assessment and again post-intervention (an expected average of 6 weeks later)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 6 Week Aerobic Exercise Intervention: Participants randomly assigned to the exercise condition will complete an 18 session aerobic exercise manipulation supervised by an American College of Sports Medicine-certified personal trainer (3 exercise sessions per week for 6 weeks).Immediately before and after participating in this intervention arm, participants will undergo the placebo-controlled morphine and naloxone administration intervention to assess mechanisms of exercise-related changes.
  exercise: Each exercise session will consist of a 5 minute warm-up, 30 minutes of aerobic exercise, followed by a 5 minute cool-down period. Aerobic exercise will consist of treadmill walking/running, stepping, elliptical, or cycling exercise as preferred by the participant. Duration of exercise will be standardized at 30 minutes with a target exercise intensity between 70-85% Heart Rate Reserve (RPE = 15, hard). Because of the focus on de-conditioned individuals with Chronic Low Back Pain, the duration and intensity of exercise will
- Normal Exercise (Control): Participants assigned to the control condition will not undergo any manipulation during this 6 week period, and will be asked to continue their current activity levels and not engage in any additional exercise activity during the study period. Immediately before and after participating in this intervention arm, participants will undergo the placebo-controlled morphine and naloxone administration intervention to assess mechanisms of exercise-related changes.
  Placebo: In randomized order (crossover) across 3 laboratory sessions each approximately 5 days apart, participants will receive: 1) 4 doses of saline placebo (20ml each), 2) an 8mg dose of naloxone (in 20ml saline vehicle), followed by saline, 4mg naloxone, and saline, or 3) morphine sulfate (0.03 mg/kg in 20ml saline vehicle initially, followed by 3 incremental doses of 0.02mg/kg each)
  Morphine: In randomized order (crossover) across 3 laboratory sessions each approximately 5 days apart, participants will receive: 1) 4 doses
Arm/Group | 6 Week Aerobic Exercise Intervention | Normal Exercise (Control)
Number analyzed (Participants) | 38 | 44
units on a scale
  Baseline (pre intervention) | 10.23 (9.17) | 7.83 (6.11)
  Change after 6 week intervention period | 0.45 (3.99) | -2.14 (4.61)
Statistical Analysis 1: Comparison: 6 Week Aerobic Exercise Intervention vs Normal Exercise (Control); Statistical analysis applies to change after 6 week intervention period; Test type: Superiority; p = .03, ANCOVA

4. Secondary Outcome: Mean Within-participant Changes From Pre- to Post-intervention in Opioid Blockade Effects (Within-participant Difference Between Naloxone and Placebo Conditions) for Ratings of Acute Thermal Pain Intensity on the McGill Pain Questionnaire-Short Form
Description: Between-participant (aerobic exercise vs. control group) comparison of mean changes from pre- to post-intervention in opioid blockade effects for ratings of acute thermal pain intensity on the McGill Pain Questionnaire-Short Form based on 3 laboratory testing days at baseline (pre-intervention) and post intervention. The score ranges from 0-33 where 0 represents no pain and 33 represents more intense pain. Positive values indicate increased endogenous opioid analgesia post intervention.
  This measure will test for endogenous opioid mechanisms of the exercise (versus control) intervention as indexed by changes in opioid blockade effects (the difference in laboratory evoked pain response evoked between placebo and naloxone drug conditions).
  This is a mixed within-between subject design. Per the study protocol, the intent of outcome measures 4 and 6 was to capture opioid blockade effects (within-participant placebo-naloxone condition difference scores) at both the pre- and post-in
Time Frame: At pre-intervention baseline laboratory assessment and again post-intervention (an expected average of 6 weeks later)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 6 Week Aerobic Exercise Intervention: Participants randomly assigned to the exercise condition will complete an 18 session aerobic exercise manipulation supervised by American College of Sports Medicine-certified personal trainer (3 exercise sessions per week for 6 weeks). Immediately before and after participating in this intervention arm, participants will undergo the placebo-controlled morphine and naloxone administration intervention to assess mechanisms of exercise related changes.
  exercise: Each exercise session will consist of a 5 minute warm-up, 30 minutes of aerobic exercise, followed by a 5 minute cool-down period. Aerobic exercise will consist of treadmill walking/running, stepping, elliptical, or cycling exercise as preferred by the participant. Duration of exercise will be standardized at 30 minutes with a target exercise intensity between 70-85% Heart Rate Reserve (RPE = 15, hard). Because of the focus on de-conditioned individuals with Chronic Low Back Pain, the duration and intensity of exercise wil
Arm/Group | 6 Week Aerobic Exercise Intervention | Normal Exercise (Control)
Number analyzed (Participants) | 38 | 44
units on a scale
  Baseline (pre intervention) | -0.33 (4.55) | 0.92 (3.81)
  Change after 6 week intervention period | 1.97 (6.32) | -0.61 (5.81)
Statistical Analysis 1: Comparison: 6 Week Aerobic Exercise Intervention vs Normal Exercise (Control); Statistical analysis applies to change after 6 week intervention period; Test type: Superiority; p = 0.17, ANCOVA

5. Secondary Outcome: Mean Change in McGill Pain Questionnaire-2 Total Chronic Back Pain Ratings
Description: Mean change in McGill Pain Questionnaire-2 total chronic back pain ratings on 3 testing days at baseline (pre intervention) and post intervention. The score ranges from 0-10 where 0 represents no pain and 10 represents most intense pain. Positive values indicate decreased back pain post intervention.
Time Frame: At pre-intervention baseline laboratory assessment and again post-intervention (an expected average of 6 weeks later)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 6 Week Aerobic Exercise Intervention | Normal Exercise (Control)
Number analyzed (Participants) | 38 | 44
units on a scale
  Baseline (pre intervention) | 2.66 (1.65) | 3.01 (1.78)
  Change after 6 week intervention period | 1.60 (1.58) | 1.36 (1.41)
Statistical Analysis 1: Comparison: 6 Week Aerobic Exercise Intervention vs Normal Exercise (Control); Statistical analysis applies to change after 6 week intervention period; Test type: Superiority; p = 0.13, ANCOVA

6. Secondary Outcome: Mean Within-participant Changes From Pre- to Post-intervention in Opioid Blockade Effects (Within-participant Difference Between Naloxone and Placebo Conditions) for McGill Pain Questionnaire-2 Total Ratings of Back Pain.
Description: Between-participant (aerobic exercise vs. control group) comparison of mean changes from pre- to post-intervention in opioid blockade effects for McGill Pain Questionnaire-2 Total ratings of back pain based on 3 laboratory testing days at baseline (pre intervention) and post intervention. The score ranges from 0-10 where 0 represents no pain and 10 represents most intense pain. Positive values indicate increased endogenous opioid analgesia post intervention.
  This measure will test the effects of the exercise (versus control) intervention on clinical outcomes as indexed by changes in opioid blockade effects (the difference in laboratory evoked pain response evoked between placebo and naloxone drug conditions).
  This is a mixed within-between subject design. Per the study protocol, the intent of outcome measures 4 and 6 was to capture opioid blockade effects (within-participant placebo-naloxone condition difference scores) at both the pre- and post-intervention lab assessments, an
Time Frame: At pre-intervention baseline laboratory assessment and again post-intervention (an expected average of 6 weeks later)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 6 Week Aerobic Exercise Intervention | Normal Exercise (Control)
Number analyzed (Participants) | 38 | 44
units on a scale
  Baseline (pre intervention) | 0.11 (0.82) | 0.18 (0.69)
  Change after 6 week intervention period | -0.12 (0.96) | -0.24 (1.28)
Statistical Analysis 1: Comparison: 6 Week Aerobic Exercise Intervention vs Normal Exercise (Control); Statistical analysis applies to change after 6 week intervention period; Test type: Superiority; p = .98, ANCOVA

7. Secondary Outcome: Mean Change in Positive and Negative Affect Scale-Negative Affect Subscale Ratings.
Description: Mean change in Positive and Negative Affect Scale-Negative Affect subscale ratings on 3 testing days at baseline (pre intervention) and post intervention. . Scale ratings range from 10 to 50 where 10 represents lowest negative affect possible and 50 represents highest negative affect possible. Positive values indicate decreased negative affect post intervention.
Time Frame: At pre intervention baseline and again post-intervention (an expected average of 6 weeks later)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 6 Week Aerobic Exercise Intervention | Normal Exercise (Control)
Number analyzed (Participants) | 38 | 44
units on a scale
  Baseline (pre intervention) | 16.38 (5.85) | 15.43 (4.52)
  Change after 6 week intervention period | 0.45 (3.99) | -2.14 (4.61)
Statistical Analysis 1: Comparison: 6 Week Aerobic Exercise Intervention vs Normal Exercise (Control); Statistical analysis applies to change after 6 week intervention period; Test type: Superiority; p = 0.52, ANCOVA

8. Secondary Outcome: Mean Change in Morphine Condition Visual Analog Scale (VAS) Opioid Effects Scale-Euphoria Subscale Ratings
Description: Mean change in morphine condition VAS Opioid Effects-Euphoria subscale ratings on 3 testing days at baseline (pre intervention) and post intervention. The score ranges from 0-300 where 0 means no euphoria and 300 means most euphoria possible. Positive values indicate decreased euphoria post intervention.
Time Frame: At pre-intervention baseline and again post-intervention (an expected average of 6 weeks later)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 6 Week Aerobic Exercise Intervention | Normal Exercise (Control)
Number analyzed (Participants) | 38 | 44
units on a scale
  Baseline (pre intervention) | 100.60 (70.35) | 108.24 (81.27)
  Change after 6 week intervention period | 3.19 (47.91) | 0.75 (50.17)
Statistical Analysis 1: Comparison: 6 Week Aerobic Exercise Intervention vs Normal Exercise (Control); Statistical analysis applies to change after 6 week intervention period; Test type: Superiority; p = 0.65, ANCOVA

9. Secondary Outcome: Mean Change in Morphine Condition Visual Analog Scale (VAS) Opioid Effects Scale-Sedation Subscale Ratings
Description: Mean change in morphine condition VAS Opioid Effects-Sedation subscale ratings on 3 testing days at baseline (pre intervention) and post intervention. The score ranges from 0-300 where 0 means no sedation and 300 means most sedation possible. Positive values indicate decreased sedation post intervention.
Time Frame: At pre-intervention baseline and again post-intervention (an expected average of 6 weeks later)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 6 Week Aerobic Exercise Intervention | Normal Exercise (Control)
Number analyzed (Participants) | 38 | 44
units on a scale
  Baseline (pre intervention) | 66.58 (71.54) | 30.63 (53.54)
  Change after 6 week intervention period | 12.89 (55.30) | -9.95 (38.033)
Statistical Analysis 1: Comparison: 6 Week Aerobic Exercise Intervention vs Normal Exercise (Control); Statistical analysis applies to change after 6 week intervention period; Test type: Superiority; p = 0.1, ANCOVA

10. Secondary Outcome: Mean Change in Morphine Condition Visual Analog Scale (VAS) Opioid Effects - Unpleasantness Subscale Ratings
Description: Mean change in morphine condition VAS Opioid Effects - Unpleasantness subscale ratings on 3 testing days at baseline (pre intervention) and post intervention. The score ranges from 0-300 where 0 represents no unpleasantness and 300 represents most unpleasantness possible. Positive values indicate decreased unpleasantness post intervention.
Time Frame: At pre-intervention baseline and again post-intervention (an expected average of 6 weeks later)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 6 Week Aerobic Exercise Intervention | Normal Exercise (Control)
Number analyzed (Participants) | 38 | 44
units on a scale
  Baseline (pre intervention) | 33.58 (36.33) | 16.52 (24.95)
  Change after 6 week intervention period | -3.21 (38.43) | 1.86 (17.99)
Statistical Analysis 1: Comparison: 6 Week Aerobic Exercise Intervention vs Normal Exercise (Control); Statistical analysis applies to change after 6 week intervention period; Test type: Superiority; p = .046, ANCOVA

11. Secondary Outcome: Mean Change in Morphine Condition Drug Effects, Liking, and Take Again (DELTA) -Drug Effect Subscale Ratings
Description: Mean change in morphine condition Drug Effects, Liking, and Take Again (DELTA) -Drug Effect subscale ratings on 3 testing days at baseline (pre intervention) and post intervention. The score ranges from 1-5 where 1 represents no effect and 5 represents very strong effect. Positive values indicate decreased overall drug effects post intervention.
Time Frame: At pre-intervention baseline and again post-intervention (an expected average of 6 weeks later)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 6 Week Aerobic Exercise Intervention: Participants randomly assigned to the exercise condition will complete an 18 session aerobic exercise manipulation supervised by an American College of Sports Medicine certified personal trainer (3 exercise sessions per week for 6 weeks). Immediately before and after participating in this intervention arm, participants will undergo the placebo-controlled morphine and naloxone administration intervention to assess mechanisms of exercise-related changes.
  exercise: Each exercise session will consist of a 5 minute warm-up, 30 minutes of aerobic exercise, followed by a 5 minute cool-down period. Aerobic exercise will consist of treadmill walking/running, stepping, elliptical, or cycling exercise as preferred by the participant. Duration of exercise will be standardized at 30 minutes with a target exercise intensity between 70-85% Heart Rate Reserve (RPE = 15, hard). Because of the focus on de-conditioned individuals with Chronic Low Back Pain, the duration and intensity of exercise wil
Arm/Group | 6 Week Aerobic Exercise Intervention | Normal Exercise (Control)
Number analyzed (Participants) | 38 | 44
units on a scale
  Baseline (pre intervention) | 2.72 (0.99) | 2.52 (1.00)
  Change after 6 week intervention period | 0.10 (1.19) | -0.12 (0.79)
Statistical Analysis 1: Comparison: 6 Week Aerobic Exercise Intervention vs Normal Exercise (Control); Statistical analysis applies to change after 6 week intervention period; Test type: Superiority; p = 0.61, ANCOVA

12. Secondary Outcome: Mean Change in Morphine Condition Drug Effects, Liking, and Take Again (DELTA) -Drug Liking Subscale Ratings
Description: Mean change in morphine condition Drug Effects, Liking, and Take Again (DELTA) -Drug Liking subscale ratings on 3 testing days at baseline (pre intervention) and post intervention. The score ranges from 0-100 where 0 represents dislike a lot and 100 represents like a lot. Positive values indicate decreased drug liking post intervention.
Time Frame: At pre-intervention baseline and again post-intervention (an expected average of 6 weeks later)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 6 Week Aerobic Exercise Intervention | Normal Exercise (Control)
Number analyzed (Participants) | 38 | 44
units on a scale
  Baseline (pre intervention) | 52.03 (12.52) | 52.89 (17.57)
  Change after 6 week intervention period | 4.13 (15.50) | 1.04 (18.68)
Statistical Analysis 1: Comparison: 6 Week Aerobic Exercise Intervention vs Normal Exercise (Control); Statistical analysis applies to change after 6 week intervention period; Test type: Superiority; p = 0.4, ANCOVA

13. Secondary Outcome: Mean Change in Morphine Condition Drug Effects, Liking, and Take Again (DELTA) -Take Again Subscale Ratings
Description: Mean change in morphine condition Drug Effects, Liking, and Take Again (DELTA) -Take Again subscale ratings on 3 testing days at baseline (pre intervention) and post intervention. The score ranges from 0-100 where 0 represents definitely would not take again and 100 represents definitely would take again. Positive values indicate decreased desire to take the drug again post intervention.
Time Frame: At pre-intervention baseline and again post-intervention (an expected average of 6 weeks later)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 6 Week Aerobic Exercise Intervention | Normal Exercise (Control)
Number analyzed (Participants) | 38 | 44
units on a scale
  Baseline (pre intervention) | 54.49 (14.54) | 55.04 (22.93)
  Change after 6 week intervention period | 4.40 (19.72) | 1.70 (22.56)
Statistical Analysis 1: Comparison: 6 Week Aerobic Exercise Intervention vs Normal Exercise (Control); Statistical analysis applies to change after 6 week intervention period; Test type: Superiority; p = 0.57, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from consent to the completion of the last study visit.(approximately 12 weeks).
Arm/Group | Exercise Plus Placebo/Morphine/Naloxone | Placebo/Morphine/Naloxone
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/44
Other Adverse Events (participants affected / at risk) | 0/38 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT02469077/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2015-07-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT02469077/Prot_SAP_001.pdf